CLINICAL TRIAL: NCT03045510
Title: A Single-center Prospective Clinical Trial of the Efficacy and Safety of Ultra Small Dose Decitabine for the Lower Risk Myelodysplastic Syndrome Patients With Transfusion Dependent
Brief Title: Efficacy and Safety of Ultra Small Dose Decitabine for the Lower Risk MDS Patients With Transfusion Dependent
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shandong University (Other)
Responsible Party: Principal Investigator, Ming Hou, Professor and Director, Shandong University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: lower risk MDS-decitabine
Record Dates: First submitted 2017-02-03; First posted 2017-02-07 (Estimated); Last update posted 2017-02-07 (Estimated); Status verified 2017-01

CONDITIONS: Myelodysplastic Syndromes
Keywords: Decitabine Myelodysplastic syndrome
MeSH Terms: conditions — Myelodysplastic Syndromes | interventions — Decitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Ultra small dose decitabine (Experimental): Decitabine 3.5mg/m2，ivdrip，qd x 5d, every four weeks for one cycle. It will be given six cycles.
  Interventions: Drug: decitabine

INTERVENTIONS:
Drug: decitabine — Decitabine 3.5mg/m2，ivdrip，qd x 5d, every four weeks for one cycle. It will be given six cycles.
  Other Names: ultra small dose decitabine

SUMMARY:
Myelodysplastic syndrome (MDS) is widely recognized as a clonal hematopoietic stem cell disorder. Decitabine has been approved for the treatment of all subtypes of myelodysplastic syndrome (MDS). However, the use of decitabine is often limited by its severe toxicity represented by myelosuppression even at relatively low doses. In lower-risk patients (including IPSS low and int-1 risk groups), treatment mainly aims at improving cytopenias, especially anemia. However, although several drugs may improve anemia, sometimes durably, most of lower risk MDS eventually require red blood cell (RBC) transfusions during their disease course. Long term RBC transfusions lead to iron overload mainly due to an increase in reticulo-endothelial iron recycling.Cardiac, liver and endocrine (diabetes mellitus) dysfunction due to iron overload and often leading to fatal outcome has been reported in heavily transfused lower risk MDS patients.

To date, the optimal regimen for decitabine treatment is not well established. In this study, we perform a prospective analysis to explore the decitabine schedule for the treatment of lower risk myelodysplastic syndrome patients with transfusion dependent.

DETAILED DESCRIPTION:
The investigators are undertaking a single-center, single-arm study of 50 lower risk myelodysplastic syndrome patients with transfusion dependent from Shandong University Qilu Hospital . All the participants are selected to receive ultra small dose decitabine treatment (given intravenously at a dose of 3.5mg/m2, qd x 5d, every four weeks for one cycle). A routine blood examination is performed twice every week. Bone marrow (BM) is examined with routine aspirate smear and G-banding analysis every 1-2 treatment courses to evaluate responses.Adverse events are also recorded throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of MDS
* The IPSS [17] score ≤ 1
* patients with transfusion dependent
* Adequate hepatic and renal function (aspartate aminotransferase [AST] ≤ 2.5 x upper normal limit, alanine aminotransferase [ALT] ≤ 2.5 x upper normal limit, bilirubin ≤ 1.5 x upper normal limit and creatinine < 2 x upper normal limit, Ccr > 60ml/min ).

Exclusion Criteria:

* Decitabine and Arsenic trioxide allergy
* Pregnancy and lactation
* Cardiovascular disease
* ECOG score > 2
* HCV, HIV, HBsAg seropositive status

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2016-12-01 (Actual); Primary Completion 2018-12-30 (Estimated); Study Completion 2020-07-30 (Estimated)

PRIMARY OUTCOMES:
complete response | 30 days from the emrollment
  Bone marrow blasts not more than 5%, absolute neutrophil count more than 1*10^9/L, HgB more than 100g/L, and platelet count more than 100*10^9/L.

CONTACTS AND LOCATIONS:
Overall Officials: Ming Lv, Doctor, Principal Investigator — Shandong University
Locations (2):
- China (2):
  - Qilu hospital, Shandong University, Jinan, Shandong
  - Shandong University Qilu Hospital, Jinan, Shandong

IPD SHARING:
Plan to Share IPD: Undecided